CLINICAL TRIAL: NCT06819098
Title: Adapted Multicomponent Training (Adapted Physical and Sports Activity - APA) for Promoting Well-being in Individuals Already Affected by Cardiovascular Diseases in Currently Stable or Chronic Conditions
Brief Title: Comparing Multicomponent and Isometric Multicomponent Training: Impact on Fitness, Health, and Life Quality in Heart Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Luca Poli, Dr., University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0324885
Record Dates: First submitted 2025-01-22; First posted 2025-02-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases
Keywords: Blood pressure; Physical activity; Resistance training; Isometric training; Health status; Quality of life
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multicomponent Training (MCT) (Experimental): subjects assigned to the MCT group will perform a training protocol defined multicomponent training, which includes aerobic, resistance and flexibility components.
  Interventions: Other: Multicomponent Training Protocol
- Isometric Multicomponent Training (IMCT) (Experimental): subjects assigned to the IMCT group will perform the same training protocol of MCT group but resistance training componet will be replaced with isometric one.
  Interventions: Other: Isometric Multicomponent Training
- Waiting List Control Group (WLCG) (No Intervention): Subjects assigned to the WLCG group will not engage in any structured physical activity throughout the intervention period, continuing with their usual lifestyle, and will be placed on a waiting list, ensuring their participation in adapted physical activity at the end of the 24-week intervention.

INTERVENTIONS:
Other: Multicomponent Training Protocol — Each session consists of:
  Warm-up (10 minutes): Low-intensity walking (Borg scale 10-11) to increase heart rate, improve blood flow, and prepare joints.
  Main phase (40 minutes):
  Aerobic exercises: Controlled jumping jacks, step-ups, alternating knee lifts, lateral steps, and leg lifts.
  Mobility exercises: Thoracic extensions, cat-to-cows, overhead stretching with a stick, and hip internal rotations (1-3 sets, 30-60 seconds per exercise).
  Resistance training: Gradual progression of 8 exercises targeting major muscle groups, such as squats, bicep curls, shoulder presses, and rows (1-3 sets, 10-15 reps, RPE 13-15).
  Cool-down (10 minutes): Breathing exercises and stretching (1-3 sets, 10-30 seconds per stretch).
  Arms: Multicomponent Training (MCT)
Other: Isometric Multicomponent Training — Each session consists of:
  Warm-up (10 minutes): Low-intensity walking (Borg scale 10-11) to increase heart rate, improve blood flow, and prepare joints.
  Main phase (40 minutes):
  Aerobic exercises: Controlled jumping jacks, step-ups, alternating knee lifts, lateral steps, and leg lifts.
  Mobility exercises: Thoracic extensions, cat-to-cows, overhead stretching with a stick, and hip internal rotations (1-3 sets, 30-60 seconds per exercise).
  Isometric training: Gradual progression of 8 isometric exercises targeting major muscle groups, such as wall squats, isometric bicep curls, lateral raises, and rows (1-3 sets, 30 seconds per exercise, RPE 13-15).
  Cool-down (10 minutes): Breathing exercises and stretching (1-3 sets, 10-30 seconds per stretch).
  Arms: Isometric Multicomponent Training (IMCT)

SUMMARY:
The goal of this clinical trial is to evaluate if a multicomponent training program (MCT), including aerobic and resistance exercises, or an isometric multicomponent training program (IMCT) can improve physiological, physical fitness, mental well-being, and quality of life in adults and elderly with a history of cardiovascular diseases (CVDs) currently stabilized. The main questions it aims to answer are:

Does MCT or IMCT improve physiological parameters, physical fitness, mental well-being, and overall quality of life compared to a waitlist control group (WLCG)? Does IMCT provide superior physiological improvements compared to MCT?

Researchers will compare:

* MCT (a combination of aerobic, mobility, and resistance training exercises)
* IMCT (a combination of aerobic, mobility, and isometric exercises) to see if these interventions improve health and quality of life outcomes compared to WLCG (participants not engaging in structured physical activity during the study), and if there will be significant physiological differences between MCT and IMCT .

Participants will:

* Complete assessments of anthropometric, hemodynamic, physical fitness, and psychological parameters at baseline (T0) and after 24 weeks (T1).
* Be randomly assigned to one of three groups (MCT, IMCT, or WLCG).
* Engage in a 24-week structured training program (MCT or IMCT) supervised by exercise professionals, including:
* Warm-up sessions (10 minutes, low-intensity walking).
* Main sessions (40 minutes): aerobic, mobility, resistance (MCT), or isometric (IMCT) exercises.
* Cool-down sessions (10 minutes): breathing and stretching exercises.

This study will provide insights into the efficacy of tailored physical activity interventions for individuals with a history of cardiovascular conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women/Men
* Aged 45-80 years
* Absence of severe medical conditions (unstable coronary artery disease, decompensated heart failure, severe pulmonary hypertension) or acute onset conditions that would prevent safe participation in physical activity, according to guidelines from the American College of Sports Medicine (ACSM), American Heart Association (AHA), and European Society of Cardiology (ESC).
* History of cardiovascular dysfunctions currently stabilized.
* Sedentary lifestyle (individuals who have not followed WHO guidelines for aerobic and resistance exercise in the past 3 months).

Exclusion Criteria:

* Smokers
* Expected absence of more than one week during the intervention period
* Lack of a medical certificate for non-competitive sports fitness
* Severe musculoskeletal or joint disorders with significant mobility limitations
* Presence of joint pain, dizziness, chest pain, or angina during physical activity
* High blood pressure: PBP ≥ 160/100 (untreated)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate | 24-weeks
  Measured with an average of 3 readings by an automated measurement device (bpm) resting heart rate and peripheral blood pressure (systolic and diastolic blood pressure) will be measured, using the automated oscillometric device.
Change in Resting Diastolic Blood pressure | 24-weeks
  Measured with an average of 3 readings by an automated measurement device as per the ESC guidelines (mmHg)
Change in Resting Systolic Blood pressure | 24-weeks
  Measured with an average of 3 readings by an automated measurement device as per the ESC guidelines (mmHg)
Change in lower body strength | 24-weeks
  30-s chair stand (30CST) test: Sit-to-stand from a chair during 30 seconds (measured in seconds)
Change in functional mobility | 24-weeks
  Timed Up and Go (TUG) Test (measured in seconds)
Change in Handrigp Strength | 24-weeks
  Handgrip Strength (HGS) test: muscle strength measured with manual dynamometers (Kgf)
Change in aerobic capacity | 24-weeks
  2-Minute Step Test (TMST): march in place for 2 minutes, lifting their knees to a height halfway between the iliac crest and the patella.The number of full knee lifts (repetitions) completed in 2 minutes is recorded.
Change in psychological parameters. | 24-weeks
  SF-36 (Short Form-36) questionnaire: to measure overall health-related quality of life. Scoring range from 0 to 100, where zero indicates the lowest worst health and 100 indicates the best health.

SECONDARY OUTCOMES:
Evaluation of motivation | 24-weeks
  BREQ-3 (Behavioral Regulation in Exercise Questionnaire-3): to assess individuals' motivation for exercise based on the Self-Determination Theory (SDT). Each item is rated on a Likert scale (e.g., 0 = "Not true for me" to 4 = "Very true for me"). Scores for each subscale are calculated by averaging the ratings of the items belonging to that subscale. The higher the score in a specific dimension, the stronger that type of motivation.
Evaluation of enjoyment | 24-weeks
  BREQ-3 (Behavioral Regulation in Exercise Questionnaire-3): Scores for intrinsic motivation subscale (calculated by averaging the ratings of the items belonging to that subscale) could be used as a proxy to assess the enjoyment levels. Each item is rated on a Likert scale (e.g., 0 = "Not true for me" to 4 = "Very true for me").The higher the score the stronger the outcome.
Evaluation of adherence to training protocols | 24-weeks
  Adherence (%): (Number of prescribed activities/Number of completed activities )×100

CONTACTS AND LOCATIONS:
Overall Officials: Luca Poli, Dr., Principal Investigator — University of Bari Aldo Moro
Locations (1):
- Società Ginnastica Angiulli, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT06819098/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT06819098/ICF_001.pdf